CLINICAL TRIAL: NCT06054204
Title: Lecturer of Oral &Maxillofacial Surgery
Brief Title: Retrieval of Displaced Root in the Maxillary Sinus Via Lateral Bony Window Using the Piezoelectric Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, mona samy sheta, lecturer of oral and maxillofacial surgery department, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Oroantral Fistula; Displaced Tooth
Keywords: displaced root; maxillary sinus; lateral bony window; piezoelectric device
MeSH Terms: conditions — Oroantral Fistula

STUDY DESIGN:
Intervention Model Description: single group assignment patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lateral bony window in maxillary sinus (Experimental): a displaced root in maxillary sinus which will be removed through a rectangular bony window will be done on the lateral wall of sinus using piezo-electric device after elevation of a full thickness mucoperiosteal flap, then the bony window will be repositioned, and the flap will be sutured.
  Interventions: Device: lateral bony window

INTERVENTIONS:
Device: lateral bony window — bony window will be made on lateral maxillary sinus wall using piezo-electric device after elevation of full thickness mucoperiosteal membrane

SUMMARY:
Ten patients with displaced root in maxillary sinus will be included in this study. the root will be recieved via lateral bony window in maxillary sinus wall using peizoelectric device then the bony window will be repositioned in its place.The patients will be received, clinically and radiologically examined, managed and followed up at the Oral and Maxillofacial surgery Department, Faculty of Dentistry, Tanta University

DETAILED DESCRIPTION:
Purpose: This study is designed to allow removal of displaced root from maxillary sinus with minimal surgical injury and simultaneous preservation of the integrity of the lateral wall of maxillary sinus by repositioning of osteotomized lateral bony window.

Materials & Methods: Ten patients with displaced root in maxillary sinus will be included in this study.

surgical procedure: A full thickness flap will be elevated to expose the lateral wall of the sinus and a rectangular bony window will be done, then the sinus lining will be incised, the displaced root will be delivered, the bony window will be repositioned, and the flap will be sutured.

Preoperative evaluation: The patients will be evaluated clinically for presence of inflammation, infection or oroantral communication and radiographically using computed tomography (CT) scan to identify the position of the displaced root.

Postoperative evaluation: The patients will be evaluated clinically each week for one month regarding to healing, presence of infection, inflammation. Radiographically, immediate panoramic view to evaluate the position of bony window and four months later to evaluate bone healing CT scan.

ELIGIBILITY:
Inclusion Criteria:

root displaced in maxillary sinus absence of infection

Exclusion Criteria:

* • patients taking medications that affect bone healing
* patients underwent head and neck radiotherapy

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
1. degree of pain evaluated clinically | one-two weeks
  using visual analogue scale:0 represent no pain and 10 represents the highest level of pain
soft tissue healing evaluated clinically | one- two week
  presence of dehiscence and exposure of bone or not
the position of bony window evaluated radiographically | one week
  using panoramic view to evaluate the precise position of bony window
bony window osteointegration and density evaluated radiographically | four months
  CT scan will be used using hounsfield units to evaluate density >1250 D1 850-1250 D2 350-850 D3 150-350 D4

SECONDARY OUTCOMES:
inflammation clinically | one week
  0 no inflammation 1-3 mild inflammation 4-7 moderate inflammation 8-10 sever inflammation 0 no inflammation 1-3 mild inflammation 4-7 moderate inflammation 8-10 sever inflammation 0 no inflammation 1-3 mild inflammation 4-7 moderate inflammation 8-10 sever inflammation

CONTACTS AND LOCATIONS:
Overall Officials: mona s sheta, lecturer, Principal Investigator — Tanta University; marwa t Ibrahim, lecturer, Principal Investigator — Tanta University
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt